CLINICAL TRIAL: NCT05880095
Title: Healthy Aging Through Time- Restricted Eating in Adults With Overweight/Obesity and Incipient Liver Disease: the ENSATI Study
Brief Title: Healthy Aging Through Time- Restricted Eating in Adults With Overweight/Obesity and Incipient Liver Disease: ENSATI
Acronym: ENSATI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); CIBER Fisiopatología de la Obesidad y la Nutrición (Unknown)
Responsible Party: Principal Investigator, Lidia Daimiel Ruiz, Principal Investigator, IMDEA Food
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMD: PI-057
Record Dates: First submitted 2023-03-16; First posted 2023-05-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Biological Aging
Keywords: Clinical trial; Time-restricted eating; Healthy aging; Epigenetics; Obesity; Precision nutrition; Autophagy; Metabolism
MeSH Terms: conditions — Intermittent Fasting; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Open, controlled, randomized, parallel groups trial
Who Masked: Outcomes Assessor
Masking Description: Intervention groups will be randomly assessed letters A, B or C. Data analists will used masked groups in the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Unrestricted Mediterranean diet (MedD) (Experimental): The aim of this group is to serve as control group. Participants will be advised to adhere to a traditional Mediterranean diet
  Interventions: Other: Unrestricted Mediterranean diet
- Energy-reduced Mediterranean diet (MedD_RC) (Experimental): The aim of this group is to allow the comparison between a traditional caloric restriction approach and a time-restricted eating program without caloric restriction.
  Interventions: Other: Energy-reduced Mediterranean diet
- Mediterranean diet with time-restricted eating (MedD_TRE) (Experimental): This is the intervention group designed to asses the main hypothesis.
  Interventions: Other: Mediterranean diet with time-restricted eating

INTERVENTIONS:
Other: Unrestricted Mediterranean diet — Participants will received nutritional educational information to encourage their adherence to a Mediterranean dietary pattern. Neither caloric restriction nor time-eating restriction will be indicated.
  Other Names: MedD
  Arms: Unrestricted Mediterranean diet (MedD)
Other: Energy-reduced Mediterranean diet — Participants will follow a Mediterranean diet with a 25% caloric restriction. Participants will be provided with dietary programs, menus, shopping lists and other educational material to encourage adherence to the intervention.
  Other Names: MEdD_RC
  Arms: Energy-reduced Mediterranean diet (MedD_RC)
Other: Mediterranean diet with time-restricted eating — Participants will follow the same dietary guidelines given to MedD group, but they must to adjust their daily meals to a self-selected 10-hour eating window. This 10h eating window of their choice should be comprised between 6.00 to 20.00h. Participants will be allowed to consume water and non-caloric drinks during the fasting period (outside the 10h eating window). Participants will be advised to follow the 10h TRE during weekdays and weekends.
  Other Names: MedD_TRE
  Arms: Mediterranean diet with time-restricted eating (MedD_TRE)

SUMMARY:
The goal of this clinical trial is to evaluate the effect of a time-restricted eating (TRE) regimen on hallmarks of aging, in comparison with traditional caloric restriction and an unrestricted diet in adults with overweight/obesity.

Investigators aim to assess:

1. If TRE is sustainable over 6-months.
2. If TRE positively affects metabolism and body composition
3. If TRE improves circadian rhythm/sleep.
4. If TRE benefits cognitive function, mood and quality of life (QoL).
5. If these beneficial effects are associated with changes in molecular hallmarks of aging.

Participants will be randomly allocated to:

* an unrestricted Mediterranean diet group (MedD)
* a energy-reduced Mediterranean diet group (MedD_RC)
* or to an unrestricted Mediterranean diet with TRE group (MedD_TRE)

Intervention will be maintained for 6 months, and there will be an additional 6-months period of follow-up to assess the maintenance of the intervention without supervision.

Changes from baseline in phenotypic and molecular hallmarks of aging, including: chronobiology, quality of life, cognition, metabolism and epigenetics among groups over the follow-up will be analyzed.

DETAILED DESCRIPTION:
Aging has been defined as the time-dependent functional decline that affects most living organisms, and this biological process occurs with great variability from person to person. Healthy aging refers to developing and maintaining functional abilities to enable the well-being of the elderly. Therefore, promoting healthy aging strategies in the population would result in people living in a healthy state for most of their lifespan. This would have an important socio-economic impact, considering that aging is a risk factor for multiple diseases and that the proportion of older persons continues to increase. Interestingly, healthy lifestyle habits such as proper nutrition and physical exercise could attenuate the progression of aging-related diseases and ameliorate age-related decline. Among the lifestyle interventions that could improve healthspan, time restricted eating (TRE) is a promising candidate. TRE is a type of intermittent fasting that involves time-limited consumption of food during a specific time window. This dietary intervention has a demonstrated positive impact on some aspects of health both in pre-clinical models and clinical trials. The beneficial effects of TRE can occur at different physiological levels that are related to healthy aging, such as metabolism and body composition, circadian rhythms and sleep, and cognitive function. However, the mechanisms through which TRE may influence these aspects are not fully understood. Therefore, and considering current evidence pointing to a beneficial effect of TRE on health, the hypothesis is that an intervention with TRE in overweight/obese individuals has a positive impact on their aging determinants (metabolism and body composition, circadian rhythms and sleep, quality of life, and cognitive function) which is associated with favorable changes in cellular traits of aging (autophagy, immunosenescence, and biological age). This is a controlled, randomized, parallel group intervention trial to assess the effect of TRE, in comparison with traditional caloric restriction and unrestricted diet on phenotypic and molecular aging parameters.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 27-35 Kg/m2
* Prevalent fatty liver disease (FLI > 59 or echography screening) EASL, Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease, 2016.
* Habitual daily eating window ≥ 14 h
* Regular sleeping patterns (7 ± 2 sleeping hours every day)
* Stable weight during the last 3 months (weight changes ≤ 4 Kg)
* Not considering changes in thei physical activity in the following 6 months
* Not being under a weight-loss program or medication.

Exclusion Criteria:

* Non-menopausal women
* Alcohol abuse (CAGE score > 2, Ewing, 1984; Malet et al. 2005)
* Change in smoking habits in the previous 6 months.
* Prevalent renal, cardiovascular, liver (excluding fatty liver), endocrine o pancreatic disease.
* Type 1 diabetes
* Type 2 diabetes with poor glucose control.
* Poorly control hypertension.
* Medical treatment affecting weight or sleep.
* Food allergies or intolerances affecting the adherence to the intervention.
* Eating disorders.
* Shift workers.
* Participants of other studies.
* Social factors affecting to the adherence to the intervention (being institutionalized, unable to ingest solid food).

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in participant's meal timing measured by questionnaires. | 12 months
  Daily time of the eating window (hours) and the daily fasting period (hours) willk be assesed through questionniares to record the meal time every day.
Change from baseline in participant's postprandial glucose levels | 12 months
  Glucose levels will be continuously monitores with glucose sensors. Glucose levels (mg/dL) 30, 60, 120 and 240 minutes after meals will be recorded.
Change from baseline in fat mass measured by bioimpedance | 12 months
  % of fat mass will be recorded by bioimpedance
Change from baseline in muscle mass measured by bioimpedance | 12 months
  % of muscle mass will be recorded by bioimpedance
Change from baseline in the blood concentration of metabolites as measured by MNR | 12 months
  MNR will be used to quantified the concentration of metabolites in blood and urine samples
Change from baseline in chronotype assessed by the morningness/eveningness (MEQ)questionnaire | 12 months
  The chronotype classification from extreme morning phenotype to extreme evening phenotype will be assessed by the MEQ questionnaires and changes in classification from baseline will be assessed
Change from baseline in sleep quality as measured with the Pittsburg's questionnaire | 12 months
  The scores obtained in Pittsburg's questionnaires in each visit will be compared with the baseline scores with mixes linear models. The score ranges from 0 to 20. Higher scores in the Pittsburg's questionnaire means worse sleeping quality.
Changes form baseline in cognitive function scores measured by the Rey Auditory Verbal Learning Test (RAVLT). | 12 months
  The scores obtained in RAVLT in each visit will be compared with the baseline scores with mixes linear models. The raw scores are corrected by age group and shown as percentil score. Higher percentile means better performance in the test.
Changes form baseline in cognitive function scores measured by STROOP color and Word test. | 12 months
  The T scores obtained in the STROOP test in each visit will be compared with the baseline scores with mixes linear models. Scores range from 20 to 80. Higher scores means better cognitive performance.
Changes from baseline in the Emotional Eating Questionnaire. | 12 months
  Changes in the classification from emotional eater to non-emotional eater will be compared among visits.
Changes from baseline in anxiety scores measured by the Hamilton Anxiety Rating Scale | 12 months
  The anxiety scores obtained in each visit will be compared with the baseline scores with mixes linear models. Higher anxiety scores means higher degree of anxiety feeling. The score ranges from 0 to 56. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. Lastly, a score of 25 to 30 indicates a moderate to severe anxiety severity.
Changes from baseline in mood scores measured by the EVEA Scale for Mood Assessment. | 12 months
  The 0-10 scores obtained in the sadness-depression, anxiety, anger/hostility and cheerfulness domains in each visit will be compared with the baseline scores with mixed linear models. Higher scores in each domains means a higher magnitude of the corresponding feeling. Scores range form 0 to 10.
Changes from baseline in health-related quality of life measured by the SF-36 questionnaire | 12 months
  The scores obtained in the different domains of the health-related quality of life questionnaire, and in the aggregated physical and mental component will be recorded and compared between visits with mixes linear models. Normalized scores range from 0 to 100 with higher scores meaning better quality of life.
Changes from baseline in well-being measured by the W-BQ12 questionnaire. | 12 months
  The total scores obtained in the well-being questionnaire in each visit will be compared with the baseline scores with mixes linear models. Scores range from 0 to 36 and higher score means better perception of well-being.
Changes from baseline in the accumulation of autophagy vacuoles | 12 months
  The dynamics of autophagy will be measured through the analysis of accumulation of autophagy vacuoles in participant's T lymphocytes and changes in the number of vacuoles comparing with baseline will be analyzed by mixed linear models.
Changes from baseline in biological age measured by the Horvath's DNAmPhenoage algorithm | 12 months
  DNA methylation will be quantified with Illumina Infinium EPIC V2.0 array and the change in methylation levels will be combined with changes in phenotypic features included in teh DNAmPhenoage algorithm. Changes comparing with baseline will be analyzed by mixed linear models.
Changes from baseline in the percentage of senescent T cells | 12 months
  Percentage of senescent T cells will be assessed by FACS using CD3 as T lymphocyte marker and CD28 as marker of senescent T cells. Percentage of senescent T cells will be calculated as the (nº of senecent T cells / Total T cells)*100. Changes from baseline will be analyzed by mixed linear models

CONTACTS AND LOCATIONS:
Locations (1):
- IMDEA Food, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Codified data and samples would be made available to other researchers upon request to the principal investigator.

REFERENCES:
- See also: Clinical trial website — https://ensati.wixsite.com/ensati
- Available data/document: Study Protocol — https://ensati.wixsite.com/ensati/qu%C3%A9-es-ensati